CLINICAL TRIAL: NCT01516333
Title: Response of Energy Peak Levels After Carbohydrates Are Eaten Glycemic Load and Satiety Study - Phase 1
Brief Title: Replace Glycemic Load and Satiety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Frank Greenway, Medial Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 26026
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Glucose Blood; Glycemic Index
Keywords: glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet 1 (Experimental): High GI; High Carb; High GL
  Interventions: Other: High GL 107
- Diet 2 (Experimental): High GI, Low Carb, Med GL
  Interventions: Other: Medium GL 76
- Diet 3 (Experimental): Low GI, High Carb, Med GL
  Interventions: Other: Medium GL 68
- Diet 4 (Experimental): Low GI, Low Carb, Low GL
  Interventions: Other: Low GL 48

INTERVENTIONS:
Other: High GL 107 — Three meals a day
  Arms: Diet 1
Other: Medium GL 76 — Three meals a day
  Arms: Diet 2
Other: Medium GL 68 — Three meals a day
  Arms: Diet 3
Other: Low GL 48 — Three meals a day
  Arms: Diet 4

SUMMARY:
The study is to examine the effect of four diets differing in glycemic index and amount of carbohydrate on blood sugar and insulin and in hunger, satiety, and vigor.

DETAILED DESCRIPTION:
The extent to which a food raises blood sugar after its consumption is ranked using the Glycemic Index (GI). Foods with a high GI are those taht cause a large and rapid rise in blood sugar while those with a low GI produce small fluctuations in blood sugar. It is believed that low GI foods are advantageous for health since the swings in blood sugar and insulin resistant or diabetic. Interestingly, some studies suggest that low GI food make you less hungry and that this may play an important role in body weight regulation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index between 25-35 kg/m2
* Fasting serum glucose
* Fasting serum glucose < 125 mg/dl
* Free of chronic disease
* Willing to eat only the foods that are provided by the Center during the diet periods
* Willing to abstain from the consumption of alcohol during the diet periods
* Regularly cycling and willing not to become pregnant using birth control (abstinence, barrier methods, partner surgically sterile
* Monophasic birth control (same dose each day)
* Hormone replacement therapy
* Post-menopausal (over 1 year without bleeding)
* Have had partial hysterectomy over the age of 55
* complete hysterectomy at any age

Exclusion Criteria:

* Documented presence of atherosclerotic disease
* Diabetes mellitus
* Renal, hepatic, endocrine, gastrointestinal, hematological or other systemic disease
* Body Mass Index <25 or > 35
* History of drug or alcohol abuse in the last year
* For women, pregnancy, breast feeding or postpartum < 6 months
* History of depression or mental illness requiring treatment or medication within that last 6 months
* Multiple food allergies or significant food preferences or restrictions that would interfere with diet adherence
* Lifestyle or schedule incompatible with the study protocol
* Planned continued use of dietary supplements through the study trial
* Smoking or tobacco use

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Blood Glucose over time | 1 month
  Blood glucose demonstrates that diets of different glycemic load result in measurable differences in serum glucose and insulin.

SECONDARY OUTCOMES:
Visual Analog scores (VAS) | 1 month
  Hunger, satiety, and vigor will be measured by the visual analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, MD, Principal Investigator — Pennington Biomedical Research Center; William Cefalu, MD, Study Chair — Pennington Biomedial Research Center; Marlene M Most, PhD, RD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Liu AG, Most MM, Brashear MM, Johnson WD, Cefalu WT, Greenway FL. Reducing the glycemic index or carbohydrate content of mixed meals reduces postprandial glycemia and insulinemia over the entire day but does not affect satiety. Diabetes Care. 2012 Aug;35(8):1633-7. doi: 10.2337/dc12-0329. Epub 2012 Jun 11. PMID 22688548